CLINICAL TRIAL: NCT00352755
Title: A Phase II Study of Surgical Debulking With Peritonectomy and Biweekly Intraperitoneal 5FU With Systemic Oxaliplatin/5FU/Leucovorin in Patients With Pseudomyxoma Peritonei or Peritoneal Carcinomatosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: after interim analysis it was determined that the risks were too great in comparision to the results
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0312
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Peritoneal Neoplasms
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Fluorouracil; Folfox protocol; Oxaliplatin; Leucovorin

ARMS (1):
- Peritonectomy + IP5FU + FOLFOX (Experimental): * Surgical debulking with peritonectomy
  * IP 5FU 600 mg/m^2 over 30-60 minutes with patient rotating every 15 minutes. Repeated every 2 weeks for a total of 9 cycles.
  * FOLFOX (oxaliplatin, 5FU, leucovorin) will follow IP therapy. Oxaliplatin 85 mg/m^2 over 2 hours with leucovorin at 400 mg/m^2 and IV 5-FU at 2400 mg/m^2 over 46 hours. Repeated every 2 weeks for a total of 8 cycles.
  Interventions: Procedure: Surgical debulking with peritonectomy; Drug: Intraperitoneal 5FU; Drug: FOLFOX

INTERVENTIONS:
Procedure: Surgical debulking with peritonectomy
Drug: Intraperitoneal 5FU
  Other Names: Fluorouracil; Efudex
Drug: FOLFOX
  Other Names: Oxaliplatin; Fluorouracil; Efudex; Leucovorin; USAN

SUMMARY:
This study prospectively evaluates a multidisciplinary approach to patients with intraperitoneal carcinomatosis at Washington University. Patients with peritoneal carcinomatosis or pseudomyxoma peritonei will undergo debulking surgery with peritonectomy and placement of adhesive barrier film followed by repeated delayed intraperitoneal chemotherapy with 5FU with systemic oxaliplatin-based chemotherapy on a biweekly schedule. A retrospective review of patients treated in a similar manner at our institution showed good tolerance and efficacy. This formal Phase II study is planned to determine the safety, toxicities and survival of patients with peritoneal carcinomatosis and pseudomyxoma peritonei treated with this regimen.

ELIGIBILITY:
Eligibility Criteria:

* Histological Diagnosis: Patients must have a histologically documented pseudomyxoma peritonei or peritoneal carcinomatosis from colorectal/appendiceal and small intestinal adenocarcinoma.
* Patients may have prior chemotherapy.
* Age: Patients must be greater than or equal to 18 years old. Because no dosing or toxicity data are currently available on the use of oxaliplatin in patients <18 years of age, children are excluded from this study, but will be eligible for other pediatric Phase I single-agent trials, when available.
* Performance Status: ECOG 0-2.
* Life Expectancy: greater than 8 weeks.
* Recovery from Intercurrent Illness: Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Hematological Status: Patients must have adequate bone marrow function defined as an absolute neutrophil count greater than or equal to 1,500/mm3, platelet count greater than or equal to 100,000/mm3 and hemoglobin greater than or equal to 8 g/dl.
* Hepatic Function: Total bilirubin must be less than or equal to institutional upper limit of normal (ULN). Transaminases (SGOT and/or SGPT) may be up to 2.5 X ULN if alkaline phosphatase is less than or equal to ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are less than or equal to ULN. However, patients who have both transaminase elevation greater than 1.5 x ULN and alkaline phosphatase greater than 2.5 x ULN are not eligible for the study.
* Renal Function: Patients must have adequate renal function defined as serum creatinine less than or equal to 2.0 mg/dl or creatinine clearance greater than or equal to 60 ml/min/1.73 m2 for patients with creatinine levels above 2.0 mg/dl.
* Sexually Active Patients: For all sexually active patients, the use of adequate barrier contraception (hormonal or barrier method of birth control) will be required during therapy, prior to study entry and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential. Pregnant and nursing women patients are not eligible.
* HIV-Positive Patients: Patients receiving anti-retroviral therapy (HAART) for HIV infection are excluded from the study because of possible pharmacokinetic interactions. Appropriate studies will be undertaken in patients receiving HAART therapy, when indicated.
* Informed Consent: After being informed of the treatment involved, patients must give written consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.
* Inclusion of Women and Minorities: Entry to this study is open to both men and women and to all racial and ethnic subgroups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Fleshman, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peritonectomy + IP5FU + FOLFOX
Started | 18
Completed | 16
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Peritonectomy + IP5FU + FOLFOX
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of the Planned Treatment Regimen as Measured by Number of Participants With Grade 3 or Higher Adverse Events
Time Frame: 30 days after end of treatment
Measure: Number; unit: participants
Arm/Group | Peritonectomy + IP5FU + FOLFOX
Number analyzed (Participants) | 18
participants
  Hemoglobin | 1
  Leukocytes | 1
  Lymphopenia | 3
  Neutrophils | 2
  Rigors/chills | 1
  Dehydration | 2
  Nausea | 3
  Vomiting | 2
  Febrile neutropenia | 1
  Anal/perianal infection | 1
  Urinary infection | 1
  Infection (clinic or micro) with Gr. 3/4 ANC | 1
  Wound infection | 2
  Alanine aminotransferase (ALT) | 1
  Creatinine | 1
  Hypermagnesemia | 1
  Hypocalcemia | 1
  Hypokalemia | 2
  Hypomagnesemia | 1
  Hyponatremia | 2
  Syncope | 1
  Abdomen pain | 3
  Head/headache pain | 1

2. Secondary Outcome: Progression Rate
Description: -Progressive disease - at least a 20% increase in the sum of the longest diameter of the target lesions taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Median follow-up was 32 months
Measure: Number; unit: percentage of participants
Arm/Group | Peritonectomy + IP5FU + FOLFOX
Number analyzed (Participants) | 16
percentage of participants | 62.5

3. Secondary Outcome: Number of Participants Who Experience Surgical Complications Associated With This Regimen
Time Frame: Median follow-up was 32 months
Measure: Number; unit: participants
Arm/Group | Peritonectomy + IP5FU + FOLFOX
Number analyzed (Participants) | 16
participants | 9

4. Secondary Outcome: Progression-free Survival
Time Frame: Median follow-up was 32 months
Measure: Median (Full Range); unit: months
Arm/Group | Peritonectomy + IP5FU + FOLFOX
Number analyzed (Participants) | 16
months | 21.20 [1.41 to 34.36]

5. Secondary Outcome: Overall Survival
Time Frame: Median follow-up was 32 months
Measure: Median (Full Range); unit: months
Arm/Group | Peritonectomy + IP5FU + FOLFOX
Number analyzed (Participants) | 16
months | 32.01 [4.27 to 35.61]

ADVERSE EVENTS:
Groups:
- Peritonectomy + IP5FU + FOLFOX: * Surgical debulking with peritonectomy
  * IP 5FU 600 mg/m2 over 30-60 minutes with patient rotating every 15 minutes. Repeated every 2 weeks for a total of 9 cycles.
  * FOLFOX (oxaliplatin, 5FU, leucovorin) will follow IP therapy. Oxaliplatin 85 mg/m2 over 2 hours with leucovorin at 400 mg/m2 and IV 5-FU at 2400 mg/m2 over 46 hours. Repeated every 2 weeks for a total of 8 cycles.
Arm/Group | Peritonectomy + IP5FU + FOLFOX
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peritonectomy + IP5FU + FOLFOX (N=18)
Dehydration (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Infection - wound (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Rigors/chills (General disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peritonectomy + IP5FU + FOLFOX (N=18)
ALT (Investigations) | 7
AST (Investigations) | 7
Abdominal pain (Gastrointestinal disorders) | 8
Alkaline phosphatase (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Bilirubin (Investigations) | 1
Blurred vision (Eye disorders) | 1
Chest/thorax pain (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Creatinine (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 7
Febrile neutropenia (Infections and infestations) | 1
Gastrointestinal, other (Gastrointestinal disorders) | 2
Head/headache (Nervous system disorders) | 1
Hematocrit (Investigations) | 2
Hemoglobin (Blood and lymphatic system disorders) | 10
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Infection - Anal/Perianal (Infections and infestations) | 1
Infection - Kidney (Infections and infestations) | 2
Infection - Oral - Cavity, gums (Infections and infestations) | 1
Infection - Urinary (Infections and infestations) | 1
Infection with Gr.3/4 neutrophils (Infections and infestations) | 1
Injection site reaction (General disorders) | 1
Insomnia (Psychiatric disorders) | 2
Leukocytes (Investigations) | 5
Lymphopenia (Investigations) | 6
Metabolic - Other (Metabolism and nutrition disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Muscle pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Neuropathy - sensory (Nervous system disorders) | 7
Neutrophils (Investigations) | 4
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1
Oral cavity (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Phlebitis (Vascular disorders) | 1
Platelets (Investigations) | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rigors/chills (General disorders) | 2
Sexual - other (Reproductive system and breast disorders) | 2
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Thrombocytopenia (Investigations) | 1
Vaginal perforation (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1
Wound infection (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes